CLINICAL TRIAL: NCT06949852
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter, Phase III Clinical Study to Evaluate the Efficacy and Safety of Nalbuphine Versus Morphine for the Treatment of Postoperative Analgesia
Brief Title: Evaluation of Safety and Efficacy of Nalbuphine Versus Morphine for Postoperative Analgesia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yangtze River Pharmaceutical Group Jiangsu Zilong Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Organization: Yangtze River Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YZJ-NBF-YZ-2303
Record Dates: First submitted 2025-04-01; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Analgesia
MeSH Terms: interventions — Nalbuphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nalbuphine group (Experimental)
  Interventions: Drug: Nalbuphine Hydrochloride Injection
- Morphine group (Active Comparator)
  Interventions: Drug: Morphine Hydrochloride Injection

INTERVENTIONS:
Drug: Nalbuphine Hydrochloride Injection — PCIA，The lockout interval is set at 10 minutes, with no background infusion.
  Arms: Nalbuphine group
Drug: Morphine Hydrochloride Injection — PCIA，The lockout interval is set at 10 minutes, with no background infusion.
  Arms: Morphine group

SUMMARY:
Evaluation of safety and efficacy of Nalbuphine versus Morphine patient controlled intravenous analgesia (PCIA) for the treatment of postoperative analgesia

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years (inclusive), regardless of gender.
2. Weight 45-100 kg (inclusive) and BMI 18.0-30.0 kg/m² (inclusive).
3. Preoperative ASA Physical Status Class I-III.
4. Scheduled for elective general anesthesia in abdominal surgery (single incision ≥5 cm) or orthopedic surgery (limb/joint procedures); completed anesthesia recovery within 4 hours postoperatively, with NRS score ≥4, and willingness to accept protocol-defined analgesia.
5. Ability to comprehend study objectives, operate PCIA devices, and communicate effectively with investigators.
6. Female subjects must be non-pregnant, non-lactating, and agree to use contraception (including partners) for 3 months post-study.
7. Voluntary participation with signed informed consent.

Exclusion Criteria:

1. Known or suspected allergy/hypersensitivity to any component of the investigational product, other opioids, or contraindicated drugs specified in the protocol .
2. Neurological/psychiatric disorders including:

   1. Clinically significant neurological diseases (e.g., epilepsy, cognitive impairment) .
   2. History of brain injury, increased intracranial pressure, or psychiatric disorders (e.g., schizophrenia, bipolar disorder, depression, anxiety) that may interfere with safety or study assessments as judged by the investigator .
3. Cardiovascular diseases/history:

   1. Severe cardiovascular conditions (NYHA Class II or higher), myocardial infarction, angina, or severe arrhythmia within the past year .
   2. Abnormal 12-lead ECG findings during screening (e.g., sinus bradycardia ≤55 bpm, ≥Grade II AV block) deemed unsuitable by the investigator .
   3. Resting systolic blood pressure ≥160 mmHg or <90 mmHg, diastolic ≥100 mmHg pre-surgery .
   4. Intraoperative circulatory instability (e.g., hypotension, bradycardia) assessed as high-risk for trial continuation .
4. Respiratory disorders/history:

   1. Bronchial asthma, high-risk respiratory depression conditions (e.g., severe COPD ≥GOLD 3, sleep apnea syndrome) .
   2. Preoperative SpO2 <93% (room air) or intraoperative respiratory depression/ventilatory dysfunction deemed unsafe .
5. Paralytic ileus, biliary/pancreatic diseases within 12 months before screening .
6. Major surgery within 3 months prior to screening.
7. Acute/chronic non-surgical pain interfering with postoperative pain assessment .
8. Preoperative anemia: Hemoglobin <70 g/L or hematocrit <25% .
9. High bleeding risk:

   1. Congenital bleeding disorders (e.g., hemophilia) .
   2. Platelet count <0.75×LLN, PT >ULN+3s, or APTT >ULN+10s .
10. Organ dysfunction:

    1. Albumin <35 g/L (untreated) .
    2. Liver/kidney function abnormalities: TBIL/ALT/AST/ALP ≥1.5×ULN ; Creatinine ≥1.5×ULN or clinically significant renal impairment; Recent dialysis (within 28 days) .
11. Random blood glucose ≥11.1 mmol/L during screening (preoperative) .
12. Participation in other clinical trials with active treatment within 3 months before surgery .
13. Other conditions deemed unsuitable by the investigator for safety or protocol compliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Sum of Pain Intensity Difference over 0-48 hours(SPID48) | 0-48 hours
  SPID48=∑PID48×[time in hours slapsed since the previous observation], PID48 denotes the pain intensity difference at time 48 hours after the first administration relative to baseline. The pain intensity is rated using an 11-point numeric scale ranging from 0 to 10, where 0 represents "no pain" and 10 represents "the worst pain imaginable."

SECONDARY OUTCOMES:
Sum of Pain Intensity Difference over 0-12 hours(SPID12) | 0-12 hours
  SPID12=∑PID12×[time in hours slapsed since the previous observation], PID12 denotes the pain intensity difference at time 12 hours after the first administration relative to baseline. The pain intensity is rated using an 11-point numeric scale ranging from 0 to 10, where 0 represents "no pain" and 10 represents "the worst pain imaginable."
Sum of Pain Intensity Difference over 0-24 hours(SPID24) | 0-24 hours
  SPID24=∑PID24×[time in hours slapsed since the previous observation], PID24 denotes the pain intensity difference at time 24 hours after the first administration relative to baseline. The pain intensity is rated using an 11-point numeric scale ranging from 0 to 10, where 0 represents "no pain" and 10 represents "the worst pain imaginable."
Sum of Pain Intensity Difference over 0-32 hours(SPID32) | 0-32 hours
  SPID32=∑PID32×[time in hours slapsed since the previous observation], PID32 denotes the pain intensity difference at time 32 hours after the first administration relative to baseline. The pain intensity is rated using an 11-point numeric scale ranging from 0 to 10, where 0 represents "no pain" and 10 represents "the worst pain imaginable."
Total Number of PCIA Pump attempts during 0~48h | 0-48 hours
  The PCIA protocol was implemented as follows: For subjects with baseline NRS scores ≥4, investigators administered the first PCIA bolus to initiate analgesia.The exact time of investigator's first PCIA activation was recorded as D0-0h. PCIA Pump Settings: Experimental Group: 2 mg per demand dose (2 mL/dose); Control Group: 1 mg per demand dose (2 mL/dose); Lockout Interval: 10 minutes. Background Infusion: None. Subsequent Analgesia Management: Following initial activation, subjects self-administered additional PCIA doses as needed based on pain levels. Subsequent PCIA Use: Subjects self-administer additional PCIA doses as needed based on pain levels. PCIA Discontinuation & Data Collection: At 48 hours (±20 min) after the first study drug administration (or upon early withdrawal), study staff will: pause and disconnect the PCIA pump, Record: total number of PCIA presses, number of effective presses and total dosage of study drug delivered via PCIA
Number of Effective Deliveries during 0~48h | 0-48 hours
  The PCIA protocol was implemented as follows: For subjects with baseline NRS scores ≥4, investigators administered the first PCIA bolus to initiate analgesia.The exact time of investigator's first PCIA activation was recorded as D0-0h. PCIA Pump Settings: Experimental Group: 2 mg per demand dose (2 mL/dose); Control Group: 1 mg per demand dose (2 mL/dose); Lockout Interval: 10 minutes. Background Infusion: None. Subsequent Analgesia Management: Following initial activation, subjects self-administered additional PCIA doses as needed based on pain levels. Subsequent PCIA Use: Subjects self-administer additional PCIA doses as needed based on pain levels. PCIA Discontinuation & Data Collection: At 48 hours (±20 min) after the first study drug administration (or upon early withdrawal), study staff will: pause and disconnect the PCIA pump, Record: total number of PCIA presses, number of effective presses and total dosage of study drug delivered via PCIA
Total Delivered Dose during 0~48h | 0-48 hours
  The PCIA protocol was implemented as follows: For subjects with baseline NRS scores ≥4, investigators administered the first PCIA bolus to initiate analgesia.The exact time of investigator's first PCIA activation was recorded as D0-0h. PCIA Pump Settings: Experimental Group: 2 mg per demand dose (2 mL/dose); Control Group: 1 mg per demand dose (2 mL/dose); Lockout Interval: 10 minutes. Background Infusion: None. Subsequent Analgesia Management: Following initial activation, subjects self-administered additional PCIA doses as needed based on pain levels. Subsequent PCIA Use: Subjects self-administer additional PCIA doses as needed based on pain levels. PCIA Discontinuation & Data Collection: At 48 hours (±20 min) after the first study drug administration (or upon early withdrawal), study staff will: pause and disconnect the PCIA pump, Record: total number of PCIA presses, number of effective presses and total dosage of study drug delivered via PCIA
Time to First Use of Rescue Medication | 0-48 hours
  Time to first use of rescue medication during 0~48h.(For subjects with inadequate pain control (NRS score ≥4) who consent to rescue therapy, the following conditions must be met before administering rescue medication: 1) NRS score remains ≥4 within 5 minutes prior to rescue drug administration; 2) At least 5 minutes have elapsed since the last effective PCIA pump press, and the next PCIA bolus is not yet due)
Proportion of Subjects Requiring Rescue Medication | 0-48 hours
Number of Rescue Medication Administrations | 0-48 hours
Proportion of Subjects with Treatment Failure | 0-48 hours
Patient Global Impression of Change (PGIC) at 48 Hours Post-Dose | 0-48 hours
  The PGIC scale (6-point) will be administered at 48h (±30min) post-dose to evaluate patients' perceived change in analgesia, ranging from 'Very much improved' (1) to 'Much worse' (6).

CONTACTS AND LOCATIONS:
Locations (24):
- China (24):
  - Peking University First Hospital, Beijing
  - Cangzhou People's Hospital, Cangzhou
  - The First People's Hospital of Changde City, Changde
  - The Third Xiangya Hospital of Central South Univerdity, Changsha
  - Heping Hospital affiliated to Changzhi Medical College, Changzhi
  - Chengdu Fifth People's Hospital, Chengdu
  - Sichuan Provincial People's Hospital, Chengdu
  - Chongqing University Affiliated Fuling Central Hospital, Chongqing
  - Deyang People's Hospital, Deyang
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - The First Affiliated Hospital of Jinan University, Guangzhou
  - The First Affiliated Hospital Of University Of South China, Hengyang
  - The Second Affiliated Hospital of Jiaxing University, Jiaxing
  - The First People's Hospital of Lianyungang, Lianyungang
  - Liuzhou Worker's Hospital, Liuchow
  - Mianyang Central Hospital, Mianyang
  - Nanjing Drum Tower Hospital, Nanjing
  - The Second Nanning People's Hospital, Nanning
  - Ningbo Medical Center LIHUILI Hospital, Ningbo
  - Ningbo NO.2 Hospital, Ningbo
  - Shanxi Bethune Hospital, Taiyuan
  - The First Affiliated Hospital of Wannan Medical College, Wuhu
  - Affiliated Hospital of Jiangnan University, Wuxi
  - Xi'an Honghui Hospital, Xi'an